CLINICAL TRIAL: NCT01978444
Title: Prospective Randomized Controlled Trial of Laparoscopic D2 Lymphadenectomy Plus Complete Mesogastrium Excision（D2+CME）vs. Laparoscopic D2 Lymphadenectomy for Advanced Gastric Cancer
Brief Title: Study on Laparoscopic D2 Lymphadenectomy Plus Complete Mesogastrium Excision（D2+CME）for Advanced Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jianping Gong, Director of Department of General Surgery, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TJ-20131101
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Gastric Cancer
Keywords: D2 lymphadenectomy; Complete Mesogastrium Excision
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: In this trial, patients and the follow-up staff are masked to the treatment allocation.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laparoscopic D2 lymphadenectomy plus CME (Experimental): Laparoscopic D2 lymphadenectomy plus CME will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Laparoscopic D2 lymphadenectomy plus CME
- laparoscopic D2 lymphadenectomy (Active Comparator): Laparoscopic D2 lymphadenectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Laparoscopic D2 lymphadenectomy

INTERVENTIONS:
Procedure: Laparoscopic D2 lymphadenectomy plus CME
  Arms: laparoscopic D2 lymphadenectomy plus CME
Procedure: Laparoscopic D2 lymphadenectomy
  Arms: laparoscopic D2 lymphadenectomy

SUMMARY:
Radical gastrectomy for gastric cancer with D2 lymph node dissection has been widely applied in advanced gastric cancer. However,for most patients,tumor local-regional recurrence has been proven unavoidable.

Recently, many clinical studies have proved that some cancer cells and cancer nodes exist in the mesogastrium which can be hardly removed by conventional radical gastrectomy with D2 lymphadenectomy. It is suggested that Complete mesogastrium excision (CME) is imperative and should be added to D2 lymphadenectomy in order to reduce the risk of local recurrence.

Thus, the comparison of short-term and long-term outcome between laparoscopic D2 lymphadenectomy plus complete mesogastrium excision and conventional laparoscopic D2 lymphadenectomy for locally advanced gastric cancer based on a well designed randomized controlled trial is needed.

ELIGIBILITY:
Inclusion Criteria:

Age from over 18 to under 75 years Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy cT2-4a, N0-3, M0 at preoperative evaluation according to the AJCC Cancer Staging Manual Seventh Edition Expected curative resection through gastrectomy with D2 lymphadenectomy Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale ASA (American Society of Anesthesiology) score class I, II, or III Informed consent obtained from patients or their appointed agent

Exclusion Criteria:

Patients treated with neoadjuvant chemotherapy or radiation therapy; Patients with history of upper abdominal surgery; History with other severe comorbidities and cannot tolerate laparoscopic surgery, such as severe heart and lung diseases, heart function below clinical stage 2, pulmonary infection, moderate to severe COPD, chronic bronchitis, severe diabetes and / or renal insufficiency, severe hepatitis and / or function below the rank of CHILD B grade, and severe malnutrition, etc; Patients suffering from malignant diseases before the study or with other gastric malignant diseases, such as lymphoma and stromal tumors, etc.; Pregnant woman and woman during lactation; Patients with mental sickness; The patient compliance is bad or the researcher expect there will not be good patient compliance;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival | 36 months
  3-years disease-free survival of the enrolled patients

SECONDARY OUTCOMES:
Postoperative recovery course | 10 days
  Time to first ambulation, flatus, liquid diet, soft diet, and duration of hospital stay. The amount of abdominal drainage and blood transfusion are also recorded.
Morbidity and mortality | 30 days; 36 months
  The early postoperative complication and mortality are defined as the event observed within 30 days after surgery, while the time frame for late complication is the period from postoperative day 31th to the end of month 36th.
  * 3-year overall survival rate [ Time Frame: 36 months ] [ Designated as safety issue: No ]
  * 3-year recurrence pattern [ Time Frame: 36 months ] [ Designated as safety issue: No ]
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type.
3-year overall survival | 36 months
  3-years overall survival of the enrolled patients

OTHER OUTCOMES:
Postoperative intraperitoneal free cancer cell (IFCC) | within 1hour
  Positive rate of cancer cells from intraperitoneal wash samples after gastrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Gong, M.D.,Ph.D., Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Tongji Medical College in Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Background] Sasako M, Saka M, Fukagawa T, Katai H, Sano T. Surgical treatment of advanced gastric cancer: Japanese perspective. Dig Surg. 2007;24(2):101-7. doi: 10.1159/000101896. Epub 2007 Apr 19. PMID 17446702
- [Background] Wu CW, Hsiung CA, Lo SS, Hsieh MC, Chen JH, Li AF, Lui WY, Whang-Peng J. Nodal dissection for patients with gastric cancer: a randomised controlled trial. Lancet Oncol. 2006 Apr;7(4):309-15. doi: 10.1016/S1470-2045(06)70623-4. PMID 16574546
- [Background] Menges M, Hoehler T. Current strategies in systemic treatment of gastric cancer and cancer of the gastroesophageal junction. J Cancer Res Clin Oncol. 2009 Jan;135(1):29-38. doi: 10.1007/s00432-008-0425-z. Epub 2008 Jun 4. PMID 18523800
- [Background] Nakamura K, Ozaki N, Yamada T, Hata T, Sugimoto S, Hikino H, Kanazawa A, Tokuka A, Nagaoka S. Evaluation of prognostic significance in extracapsular spread of lymph node metastasis in patients with gastric cancer. Surgery. 2005 May;137(5):511-7. doi: 10.1016/j.surg.2005.01.007. PMID 15855922
- [Background] Nagatomo A, Abe N, Takeuchi H, Yanagida O, Masaki T, Mori T, Sugiyama M, Ohkura Y, Fujioka Y, Atomi Y. Microscopic cancer cell spread in gastric cancer: whole-section analysis of mesogastrium. Langenbecks Arch Surg. 2009 Jul;394(4):655-60. doi: 10.1007/s00423-008-0427-y. Epub 2008 Oct 18. PMID 18931855
- [Result] Xie D, Osaiweran H, Liu L, Wang X, Yu C, Tong Y, Hu J, Gong J. Mesogastrium: a fifth route of metastasis in gastric cancer? Med Hypotheses. 2013 Apr;80(4):498-500. doi: 10.1016/j.mehy.2012.12.020. Epub 2013 Feb 10. PMID 23403142
- [Result] Xie D, Yu C, Liu L, Osaiweran H, Gao C, Hu J, Gong J. Short-term outcomes of laparoscopic D2 lymphadenectomy with complete mesogastrium excision for advanced gastric cancer. Surg Endosc. 2016 Nov;30(11):5138-5139. doi: 10.1007/s00464-016-4847-4. Epub 2016 Mar 22. PMID 27005289
- [Result] Xie D, Gao C, Lu A, Liu L, Yu C, Hu J, Gong J. Proximal segmentation of the dorsal mesogastrium reveals new anatomical implications for laparoscopic surgery. Sci Rep. 2015 Nov 6;5:16287. doi: 10.1038/srep16287. PMID 26542081
- [Result] Xie D, Liu L, Osaiweran H, Yu C, Sheng F, Gao C, Hu J, Gong J. Detection and Characterization of Metastatic Cancer Cells in the Mesogastrium of Gastric Cancer Patients. PLoS One. 2015 Nov 13;10(11):e0142970. doi: 10.1371/journal.pone.0142970. eCollection 2015. PMID 26566136
- [Result] Shen J, Cao B, Wang Y, Xiao A, Qin J, Wu J, Yan Q, Hu Y, Yang C, Cao Z, Hu J, Yin P, Xie D, Gong J. Prospective randomized controlled trial to compare laparoscopic distal gastrectomy (D2 lymphadenectomy plus complete mesogastrium excision, D2 + CME) with conventional D2 lymphadenectomy for locally advanced gastric adenocarcinoma: study protocol for a randomized controlled trial. Trials. 2018 Aug 9;19(1):432. doi: 10.1186/s13063-018-2790-5. PMID 30092843
- [Derived] Wu Y, He F, Liu L, Jiang W, Deng J, Zhang Y, Cao Z, Xu X, Gong J. The Use of CellCollector Assay to Detect Free Cancer Cells in the Peritoneal Cavity of Colorectal Cancer Patients: An Experimental Study. Cancer Med. 2024 Nov;13(21):e70378. doi: 10.1002/cam4.70378. PMID 39503055
- [Derived] Tu J, Shao S, Qin J. The number of mesogastria containing metastatic lymph nodes predicts gastric cancer prognosis. Surgery. 2024 Sep;176(3):739-747. doi: 10.1016/j.surg.2024.05.027. Epub 2024 Jun 15. PMID 38879382
- [Derived] Xie D, Shen J, Liu L, Cao B, Xiao A, Qin J, Wu J, Yan Q, Hu Y, Yang C, Cao Z, Hu J, Yin P, Gong J. Randomized clinical trial on D2 lymphadenectomy versus D2 lymphadenectomy plus complete mesogastric excision in patients undergoing gastrectomy for cancer (DCGC01 study). Br J Surg. 2024 May 3;111(5):znae106. doi: 10.1093/bjs/znae106. PMID 38713611
- [Derived] Xie D, Shen J, Liu L, Cao B, Wang Y, Qin J, Wu J, Yan Q, Hu Y, Yang C, Cao Z, Hu J, Yin P, Gong J. Complete mesogastric excision for locally advanced gastric cancer: short-term outcomes of a randomized clinical trial. Cell Rep Med. 2021 Mar 16;2(3):100217. doi: 10.1016/j.xcrm.2021.100217. eCollection 2021 Mar 16. PMID 33763656